CLINICAL TRIAL: NCT06198465
Title: Perioperative Adebrelimab and Chemotherapy in Esophageal and Esophagogastric Junction Carcinoma: a Prospective, Open-label, Single-center Clinical Study
Brief Title: Perioperative Adebrelimab and Chemotherapy in Esophageal and Esophagogastric Junction Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJEC
Record Dates: First submitted 2023-12-13; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Adebrelimab; Esophageal Cancer; Perioperative Period
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adebrelimab combined with chemotherapy (Experimental)
  Interventions: Drug: adebrelimab,Paclitaxel,Lobaplatin,Fluorouracil

INTERVENTIONS:
Drug: adebrelimab,Paclitaxel,Lobaplatin,Fluorouracil — adebrelimab: 1200mg，D1，q3w; Paclitaxel: 50mg/m2 D1/8/15； Lobaplatin: 50mg，iv 2h，d1; Fluorouracil: 400mg/m2，bolus iv，600mg/m2，iv 22h，d1-3；

SUMMARY:
The goal of this prospective, open-label, single-center clinical study is to learn about the efficacy and safety of aderbelimab combined with chemotherapy in the perioperative treatment of esophageal and esophagogastric junction cancer. The main question it aims to answer are:prediction for pCR after perioperative adebrelimab and chemotherapy in esophageal and esophagogastric junction carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, both genders;
2. Histologically or cytological confirmed esophageal and esophagogastric junction cancer (cT3-4, anyN, M0);
3. Without prior treatments including surgery, chemotherapy, radiotherapy, and targeting treatment for esophageal and esophagogastric junction cancer;
4. According to the RECIST v1.1 standard, there must be at least 1 measurable lesion;
5. ECOG PS score 0-1;
6. Adequate organ function, and there are no serious functional abnormalities or immune deficiency diseases such as blood, heart, lung, liver, kidney, bone marrow, etc. Laboratory examinations meet the following requirements:

1) Hemoglobin ≥ 90 g/L; 2) Leukocytes ≥ 3.0x10^9/L; Absolute neutrophil count≥ 1.5x10^9/L; 3) Platelet ≥ 100x10^9/L; 4) Serum creatinine ≤1.5 ULN or creatinine clearance rate≥50 mL/min; 5) Total bilirubin ≤1.5 ULN; 6) ALT ≤2.5 ULN; AST ≤2.5 ULN; 7) Urinary protein <2+; if urine protein≥2+, 24-hour urine protein quantification shows that the protein must be ≤1g; 7. Coagulation function test:

1. INR ≤1.5 ULN;
2. APTT ≤1.5 ULN;
3. PT≤1.5ULN； 8.Previous use of anti-tumor traditional Chinese medicines, Chinese patent medicines, and immunomodulators (such as thymosin, interleukins, etc.) must be ≥ 2 weeks from the start of study medication; 9. For females of child bearing potential, a negative serum/urine pregnancy test result within 72h before study treatment. For female and male participants of reproductive potential must be willing to use adequate contraception for the course of the study until 3 months after the last dose of any of the drugs in the study; 10.Volunteered to participate in the study, signed the informed consent form; 11. Had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. Suffering from any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (hormone replacement) can be included after treatment); subjects with childhood asthma that has completely resolved and do not require any intervention in adulthood or vitiligo can be included, but subjects who require medical intervention with bronchodilators are not included;
2. People with innate or acquired immune function defects, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C positive hepatitis C antibody, and high HCV-RNA (lower detection limit of the analytical method) or combined with hepatitis B and hepatitis C co-infection; patients who have used other drugs for clinical trial research within 4 weeks before the first dose;
3. Have had clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months;
4. Such as gastrointestinal bleeding, esophageal and gastric varices with bleeding risk, bleeding gastric ulcer, or vasculitis; a gastroscopy is required during the screening period. If the gastroscopy results indicate severe gastric ulcer or the researcher determines that there is bleeding, If the risk is high, you will not be eligible; gastrointestinal perforation or gastrointestinal fistula has occurred within 6 months;
5. Suffering from uncontrolled cardiac clinical symptoms or diseases, such as (1) NYHA II or above heart failure (2) unstable angina (3) myocardial infarction within 1 year (4) poorly controlled arrhythmia;
6. The number of neutrophils in peripheral blood <1500/mm3;
7. Severe infection (e.g. requiring intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks before the first dose, or unexplained fever >38.5°C during the screening period/before the first dose;
8. Those who are known to have a history of allergies to the drug components of this regimen;
9. There may be increased risks of participation in research and study medication, or other severe, acute and chronic diseases;
10. Other conditions deemed inappropriate for inclusion by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | At time of surgery
  defined as the absence of any viable tumor at the time of surgical resection, as assessed by central and local pathology laboratory

SECONDARY OUTCOMES:
R0 resection rate | At time of surgery
  R0 resection rate
Disease-Free Survival (DFS) | up to 2 year
  Time after R0 resection to disease recurrence or death Time after R0 resection to disease recurrence or death Time after R0 resection to disease recurrence or death Time after R0 resection to disease recurrence or death
Overall Survival (OS) | up to 2 year
  defined as the time from randomization to death from any cause during the course of the study.
Number of participants with treatment-related adverse events | 6 months
  assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, the Air Force Medical University, Xi'an, Shaan'xi, China